CLINICAL TRIAL: NCT07271732
Title: Songling Xuemaikang Capsules for Cerebral Small Vessel Disease: A Randomized, Double-blind, Placebo-controlled, Multicenter Clinical Study
Brief Title: Songling Xuemaikang Capsules for Cerebral Small Vessel Disease
Acronym: SXC-CSVD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Ying Gao, Prof., Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025DZMEC-188-02
Record Dates: First submitted 2025-09-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Hypertension; Cerebral Small Vessel Diseases
MeSH Terms: conditions — Hypertension; Cerebral Small Vessel Diseases | interventions — songling xuemaikang

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Songling Xuemaikang Capsule, 3 capsules/time, tid, p.o
  Interventions: Drug: Songling Xuemaikang Capsule
- Control group (Placebo Comparator): Songling Xuemaikang Capsule placebo, 3 capsules/time, tid, p.o
  Interventions: Drug: Songling Xuemaikang Capsule Placebo

INTERVENTIONS:
Drug: Songling Xuemaikang Capsule — 3 capsules/time, tid, p.o Duration of Treatment: 1 year (12 months)
  Arms: Test group
Drug: Songling Xuemaikang Capsule Placebo — 3 capsules/time, tid, p.o Duration of Treatment: 1 year (12 months)
  Arms: Control group

SUMMARY:
Cerebral small vessel disease (CSVD) is a common age-related microvascular disease related to the slow accumulation of damage to small arteries, veins, and capillaries. Hypertension is a risk factor for cerebrovascular disease, and its damage to the vascular endothelium is one of the key contributing factors to the pathogenesis of CSVD. CSVD has an insidious onset, and patients may exhibit no clinical symptoms in the early stage. Common clinical manifestations of chronic CSVD include vascular dementia, depression, gait disturbance, and abnormalities in swallowing and urinary functions. There is currently no specific treatment for CSVD.

Existing studies have shown that Songling Xuemaikang capsule (SXC) combined with antihypertensive drugs exerted significant effects on systolic blood pressure (SBP), diastolic blood pressure (DBP), 24-hour SBP, and 24-hour DBP, while also improving symptoms of hypertension. Animal experiments have demonstrated that SXC can reduce apoptosis and alleviate cerebral ischemia-reperfusion injury, exerting neuroprotective effects. Additionally, a previously completed multicenter, randomized, double-blind, non-inferiority-designed clinical trial by the team, conducted in patients with primary hypertension, showed that SXC were non-inferior to losartan potassium in reducing diastolic blood pressure. Therefore, exploring the therapeutic potential of SXC in CSVD is highly necessary.

This project is a randomized, double-blind, placebo-controlled multicenter clinical study to investigate the clinical efficacy and safety of SXC in the treatment of hypertension with CSVD. A total of 90 subjects who met the subject screening criteria are planned to be enrolled, with 45 patients in the test group and 45 patients in the placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55-75 years (both inclusive);
2. MRI has moderate to (1) severe white matter lesions (deep Fazekas score > 1 or paraventricular Fazekas score > 2 or modified Fazekas score > 1), or (2) mild white matter hyperintensity (deep Fazekas score = 1 or paraventricular Fazekas score = 2 or modified Fazekas score = 1) combined with more than 1 lacunar infarction;
3. History of essential hypertension; Hypertension is defined as SBP consistently greater than 140 mmHg and/or DBP consistently greater than 90 mmHg, or those requiring clinical antihypertensive treatment.
4. Meeting the diagnostic criteria for hyperactivity of liver yang pattern; Hyperactivity of liver yang pattern is defined as having at least three of the following six symptoms: headache, dizziness or vertigo, irritability, flushed face, red eyes, and yellow tongue coating.
5. Functional independence in daily living (Modified Rankin Scale ≤2);
6. Voluntary participation in the study and be willing to sign the Informed Consent Form.

Exclusion Criteria:

1. Patients with acute ischemic stroke or acute intracranial hemorrhage (e.g., epidural hematoma, subdural hematoma, subarachnoid hemorrhage, intracerebral hemorrhage, etc.) or a history of cerebral infarction (non-lacunar) or intracranial hemorrhage within the past 3 months;
2. Symptomatic stenosis of the middle cerebral artery and/or internal carotid artery (stenosis rate ≥50%), or asymptomatic stenosis of the middle cerebral artery and/or internal carotid artery (stenosis rate ≥70%);
3. Untreated cerebrovascular malformations or intracranial aneurysms (diameter >3 mm);
4. Significant non-vascular white matter lesions (e.g., multiple sclerosis, adult-onset leukoencephalopathy, metabolic encephalopathy, etc.);
5. Patients with a history of cognitive impairment due to other causes (e.g., normal pressure hydrocephalus, Alzheimer's disease, Parkinson's disease, multiple sclerosis, encephalitis, etc.);
6. A history of intracranial or intramedullary surgery within the past year;
7. Severe hepatic, renal, or cardiac insufficiency (ALT or AST >2 times the upper limit of normal, or serum creatinine >1.5 times the upper limit of normal, or New York Heart Association [NYHA] functional class III or IV);
8. Severe three-vessel coronary artery disease as shown by coronary computed tomography angiography or coronary angiography within 90 days or suffering from frequent angina;
9. Refractory hyperglycemia uncontrolled by medication (fasting blood glucose >10 mmol/L, or HbA1c >8.0%);
10. Patients with severe diseases such as cancer and a life expectancy of less than 2 years;
11. Patients with psychiatric disorders that affect study medication administration and evaluation;
12. Previous allergy or intolerance to Songling Xuemaikang Capsules;
13. Contraindications to MRI examination (e.g., claustrophobia, presence of an implantable pacemaker, etc.);
14. Patients unable to comply with follow-up examinations or other study procedures due to residential location or other reasons;
15. Participation in other clinical trial projects.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the volume of white matter hyperintensities at 1 year. | 1 year
  Measure changes in the volume of white matter hyperintensities on brain MRI

SECONDARY OUTCOMES:
Change from baseline in Mini-Mental State Examination (MMSE) at 1 year; | 1 year
  Change from baseline in Mini-Mental State Examination (MMSE). Score range is 0-30. Higher score means good cognition.
Change from baseline in Hamilton Anxiety Scale (HAMA) at 1 year; | 1 year
  Change from baseline in Hamilton Anxiety Scale (HAMA).Score range is 0-56. Higher score means a more severe state of anxiety.
Change from baseline in Hamilton Depression Scale (HAMD) at 1 year; | 1 year
  Change from baseline in Hamilton Depression Scale (HAMD). Score range is 0-76. Higher score means a more severe state of anxiety.
Change from baseline in Pittsburgh Sleep Quality Index (PSQI) at 1 year; | 1 year
  Change from baseline in Pittsburgh Sleep Quality Index (PSQI) at 1 year. Score range is 0-21. Higher score means worse sleep quality.
Change from baseline in Barthel Index (BI) at 1 year; | 1 year
  Change from baseline in Barthel Index (BI). Score range is 0-100. Higher score means good physical activities of daily living.
Feasibility of recruitment and retention | 1 year
  The feasibility is defined as >95% of randomized patients retained at 1 year
Change from baseline in the symptom of hyperactivity of liver yang pattern at 1 year; | 1 year
  Change from baseline in the symptom of hyperactivity of liver yang pattern, which are headache, dizziness or vertigo, irritability, flushed face, red eyes, and yellow tongue coating. The study plans to analyze whether there are statistically significant differences in the incidence of the above six symptoms before and after treatment. On the other hand, for headache, dizziness or vertigo, irritability, if they do not resolve at follow-up time points, patient-reported outcomes (PROs) will be used to record the degree of change in patients' symptoms from baseline (expressed as a percentage, with >100% indicating symptom worsening and <100% indicating symptom relief), and statistical analysis will be carried out. For flushed face, red eyes, and yellow tongue coating, binary analysis will be performed based solely on their presence or absence.
Change from baseline in the mean 24h systolic blood pressure at 1 year; | 1 year
  Change from baseline in the mean 24h systolic blood pressure
Change from baseline in the mean 24h diastolic blood pressure at 1 year; | 1 year
  Change from baseline in the mean 24h diastolic blood pressure
Change from baseline in the mean daytime systolic blood pressure at 1 year; | 1 year
  Change from baseline in the mean daytime systolic blood pressure
Change from baseline in the mean daytime diastolic blood pressure at 1 year; | 1 year
  Change from baseline in the mean daytime diastolic blood pressure
Change from baseline in the mean nighttime systolic blood pressure at 1 year | 1 year
  Change from baseline in the mean nighttime systolic blood pressure
Change from baseline in the mean nighttime diastolic blood pressure at 1 year | 1 year
  Change from baseline in the mean nighttime diastolic blood pressure
Change from baseline in the mean 24h pulse pressure at 1year | 1 year
  Change from baseline in the mean 24h pulse pressure
Change from baseline in the blood pressure load at 1 year | 1 year
  Change from baseline in the blood pressure load
Change from baseline in the official systolic blood pressure at 1 year | 1 year
  Change from baseline in the official systolic blood pressure
Change from baseline in the official diastolic blood pressure at 1 year | 1 year
  Change from baseline in the official diastolic blood pressure
Change from baseline in the official pulse pressure at 1year | 1 year
  Change from baseline in the official pulse pressure
Change from baseline in the official blood pressure compliance rate at 1 year | 1 year
  Change from baseline in the official blood pressure compliance rate

OTHER OUTCOMES:
Numbers in new vascular events from baseline to 1 year | 1 year
  New vascular events include ischemic stroke, TIA, cerebral hemorrhage, MI, pulmonary embolism, thrombosis, peripheral arterial occlusion
Numbers in all-cause hospitalization from baseline to 1 year | 1 year
  Numbers in all-cause hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Dongzhimen Hospital, Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China